CLINICAL TRIAL: NCT01649297
Title: A Randomised, Double Blind, Placebo Controlled, Parallel Group Efficacy and Safety Study of Oral Administration of Empagliflozin Twice Daily Versus Once Daily in Two Different Daily Doses Over 16 Weeks as add-on Therapy to a Twice Daily Dosing Regimen of Metformin in Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control
Brief Title: A 16 Weeks Study on Efficacy and Safety of Two Doses of Empagliflozin (BI 10773) (Once Daily Versus Twice Daily) in Patients With Type 2 Diabetes Mellitus and Preexisting Metformin Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1276.10; 2012-000905-53 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; BID protein, human

ARMS (5):
- empagliflozin (high dose qd) (Experimental): Patients receive Empagliflozin high dose once daily
  Interventions: Drug: Placebo; Drug: Empagliflozin (high dose qd)
- empagliflozin (high dose bid) (Experimental): Patients receive Empagliflozin high dose split twice daily
  Interventions: Drug: Placebo; Drug: empagliflozin (high dose bid)
- empagliflozin (low dose qd) (Experimental): Patients receive Empagliflozin low dose once daily
  Interventions: Drug: empagliflozin (low dose qd); Drug: Placebo
- empagliflozin (low dose bid) (Experimental): Patients receive Empagliflozin low dose split twice daily
  Interventions: Drug: Placebo; Drug: empagliflozin (low dose bid)
- Placebo (Placebo Comparator): Patients receive placebo matching Empagliflozin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Patients receive placebo matching empagliflozin (low dose qd)
  Arms: empagliflozin (high dose qd)
Drug: Placebo — Patients receive placebo matching empagliflozin (low dose bid)
  Arms: Placebo
Drug: Placebo — Patients receive placebo matching Empagliflozin (high dose qd)
  Arms: empagliflozin (high dose bid)
Drug: Placebo — Patients receive placebo matching Empagliflozin (high dose qd)
  Arms: empagliflozin (low dose bid)
Drug: Placebo — Patients receive placebo matching Empagliflozin (high dose qd)
  Arms: Placebo
Drug: empagliflozin (low dose qd) — Patients receive Empagliflozin low dose once daily
  Arms: empagliflozin (low dose qd)
Drug: Placebo — Patients receive placebo matching empagliflozin (low dose qd)
  Arms: empagliflozin (low dose bid)
Drug: Placebo — Patients receive placebo matching empagliflozin (low dose bid)
  Arms: empagliflozin (low dose qd)
Drug: Placebo — Patients receive placebo matching Empagliflozin (high dose bid)
  Arms: empagliflozin (high dose qd)
Drug: Placebo — Patients receive placebo matching Empagliflozin (high dose bid)
  Arms: Placebo
Drug: Placebo — Patients receive placebo matching empagliflozin (low dose qd)
  Arms: empagliflozin (high dose bid)
Drug: Placebo — Patients receive placebo matching empagliflozin (low dose bid)
  Arms: empagliflozin (high dose qd)
Drug: Placebo — Patients receive placebo matching Empagliflozin (high dose bid)
  Arms: empagliflozin (low dose bid)
Drug: Placebo — Patients receive placebo matching empagliflozin (low dose qd)
  Arms: Placebo
Drug: Placebo — Patients receive placebo matching empagliflozin (low dose bid)
  Arms: empagliflozin (high dose bid)
Drug: Placebo — Patients receive placebo matching Empagliflozin (high dose bid)
  Arms: empagliflozin (low dose qd)
Drug: Empagliflozin (high dose qd) — Patients receive Empagliflozin high dose once daily
  Arms: empagliflozin (high dose qd)
Drug: empagliflozin (high dose bid) — Patients receive Empagliflozin high dose split twice daily
  Arms: empagliflozin (high dose bid)
Drug: Placebo — Patients receive placebo matching Empagliflozin (high dose qd)
  Arms: empagliflozin (low dose qd)
Drug: empagliflozin (low dose bid) — Patients receive Empagliflozin low dose split twice daily
  Arms: empagliflozin (low dose bid)

SUMMARY:
The aim of this study is to investigate the efficacy and safety of two doses (high and low) of empagliflozin as add-on therapy to metformin in patients with type 2 diabetes mellitus (T2DM) and insufficient glycaemic control. Both doses may be given once daily or split to a twice daily dosage. This results in 4 different dosage regimens of empagliflozin (high dose once daily or split vs. low dose once daily or split). This is done to evaluate whether a twice daily dose regimen of empagliflozin results in a loss of efficacy relative to once daily dosing when given on top of metformin background therapy.

ELIGIBILITY:
Inclusion criteria:

1. confirmed diagnosis of T2DM
2. Glycated hemoglobin (HbA1c) >=7.0 and <=10/0% at Visit 1
3. Metformin therapy (at least 1500 mg/day, BID)
4. age>=18 at Visit 1
5. body mass index <=45 kg/m2

Exclusion criteria:

1. estimated creatinine clearance rate (eCCr) <60 ml/min (Cockcroft-Gault formula) screening and/or run-in
2. a confirmed glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast during placebo run-in

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 983 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (139):
- United States (39):
  - 1276.10.11036 Boehringer Ingelheim Investigational Site, Florence, Alabama
  - 1276.10.11049 Boehringer Ingelheim Investigational Site, Jonesboro, Arkansas
  - 1276.10.11040 Boehringer Ingelheim Investigational Site, Lomita, California
  - 1276.10.11033 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1276.10.11002 Boehringer Ingelheim Investigational Site, Rancho Cucamonga, California
  - 1276.10.11050 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 1276.10.11015 Boehringer Ingelheim Investigational Site, West Hills, California
  - 1276.10.11012 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 1276.10.11047 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1276.10.11010 Boehringer Ingelheim Investigational Site, Bradenton, Florida
  - 1276.10.11005 Boehringer Ingelheim Investigational Site, Davie, Florida
  - 1276.10.11004 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1276.10.11051 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1276.10.11009 Boehringer Ingelheim Investigational Site, Oakland Park, Florida
  - 1276.10.11044 Boehringer Ingelheim Investigational Site, Palm Harbor, Florida
  - 1276.10.11030 Boehringer Ingelheim Investigational Site, Dunwoody, Georgia
  - 1276.10.11027 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1276.10.11020 Boehringer Ingelheim Investigational Site, Elwood, Indiana
  - 1276.10.11001 Boehringer Ingelheim Investigational Site, Bangor, Maine
  - 1276.10.11048 Boehringer Ingelheim Investigational Site, Sterling Heights, Michigan
  - 1276.10.11058 Boehringer Ingelheim Investigational Site, Jackson, Mississippi
  - 1276.10.11055 Boehringer Ingelheim Investigational Site, Edison, New Jersey
  - 1276.10.11011 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 1276.10.11035 Boehringer Ingelheim Investigational Site, North Myrtle Beach, North Carolina
  - 1276.10.11041 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1276.10.11018 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1276.10.11043 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1276.10.11017 Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - 1276.10.11022 Boehringer Ingelheim Investigational Site, Fleetwood, Pennsylvania
  - 1276.10.11003 Boehringer Ingelheim Investigational Site, Johnson City, Tennessee
  - 1276.10.11042 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 1276.10.11013 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1276.10.11026 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1276.10.11031 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1276.10.11034 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1276.10.11028 Boehringer Ingelheim Investigational Site, Pearland, Texas
  - 1276.10.11029 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1276.10.11016 Boehringer Ingelheim Investigational Site, Port Orchard, Washington
  - 1276.10.11024 Boehringer Ingelheim Investigational Site, Spokane, Washington
- Australia (2):
  - 1276.10.61002 Boehringer Ingelheim Investigational Site, Wollongong, New South Wales
  - 1276.10.61001 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
- Canada (10):
  - 1276.10.20008 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1276.10.20005 Boehringer Ingelheim Investigational Site, Surrey, British Columbia
  - 1276.10.20010 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1276.10.20002 Boehringer Ingelheim Investigational Site, Bathurst, New Brunswick
  - 1276.10.20001 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1276.10.20007 Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - 1276.10.20006 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1276.10.20004 Boehringer Ingelheim Investigational Site, Drummondville, Quebec
  - 1276.10.20003 Boehringer Ingelheim Investigational Site, Point Claire, Quebec
  - 1276.10.20009 Boehringer Ingelheim Investigational Site, Victoriaville, Quebec
- Estonia (4):
  - 1276.10.37203 Boehringer Ingelheim Investigational Site, Pärnu
  - 1276.10.37201 Boehringer Ingelheim Investigational Site, Tallinn
  - 1276.10.37202 Boehringer Ingelheim Investigational Site, Tallinn
  - 1276.10.37204 Boehringer Ingelheim Investigational Site, Viljandi County
- France (10):
  - 1276.10.33002 Boehringer Ingelheim Investigational Site, Aire-sur-l'Adour
  - 1276.10.33003 Boehringer Ingelheim Investigational Site, Bischheim
  - 1276.10.33009 Boehringer Ingelheim Investigational Site, Bourg-des-Comptes
  - 1276.10.33014 Boehringer Ingelheim Investigational Site, Bourges
  - 1276.10.33007 Boehringer Ingelheim Investigational Site, Broglie
  - 1276.10.33001 Boehringer Ingelheim Investigational Site, Mont-de-Marsan
  - 1276.10.33008 Boehringer Ingelheim Investigational Site, Paris
  - 1276.10.33006 Boehringer Ingelheim Investigational Site, Saint Vinecnt de Tyrosse
  - 1276.10.33011 Boehringer Ingelheim Investigational Site, Segré
  - 1276.10.33004 Boehringer Ingelheim Investigational Site, Strasbourg
- Georgia (6):
  - 1276.10.99501 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1276.10.99502 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1276.10.99503 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1276.10.99504 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1276.10.99505 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1276.10.99506 Boehringer Ingelheim Investigational Site, Tbilisi
- Germany (7):
  - 1276.10.49001 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1276.10.49006 Boehringer Ingelheim Investigational Site, Berlin
  - 1276.10.49007 Boehringer Ingelheim Investigational Site, Berlin
  - 1276.10.49005 Boehringer Ingelheim Investigational Site, Essen
  - 1276.10.49004 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1276.10.49002 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1276.10.49003 Boehringer Ingelheim Investigational Site, Rehlingen-Siersburg
- Guatemala (5):
  - 1276.10.50201 Boehringer Ingelheim Investigational Site, Guatemala Ciudad
  - 1276.10.50203 Boehringer Ingelheim Investigational Site, Guatemala Ciudad
  - 1276.10.50204 Boehringer Ingelheim Investigational Site, Guatemala Ciudad
  - 1276.10.50205 Boehringer Ingelheim Investigational Site, Guatemala Ciudad
  - 1276.10.50202 Boehringer Ingelheim Investigational Site, Quetzaltenango Ciudad
- Italy (9):
  - 1276.10.39004 Boehringer Ingelheim Investigational Site, Arenzano (GE)
  - 1276.10.39003 Boehringer Ingelheim Investigational Site, Bologna
  - 1276.10.39007 Boehringer Ingelheim Investigational Site, Catanzaro
  - 1276.10.39009 Boehringer Ingelheim Investigational Site, Catanzaro
  - 1276.10.39002 Boehringer Ingelheim Investigational Site, Napoli
  - 1276.10.39006 Boehringer Ingelheim Investigational Site, Palermo
  - 1276.10.39001 Boehringer Ingelheim Investigational Site, Roma
  - 1276.10.39008 Boehringer Ingelheim Investigational Site, Roma
  - 1276.10.39005 Boehringer Ingelheim Investigational Site, Torino
- Latvia (4):
  - 1276.10.37102 Boehringer Ingelheim Investigational Site, Daugavpils
  - 1276.10.37104 Boehringer Ingelheim Investigational Site, Ogre
  - 1276.10.37101 Boehringer Ingelheim Investigational Site, Riga
  - 1276.10.37103 Boehringer Ingelheim Investigational Site, Tukums
- Lithuania (4):
  - 1276.10.37003 Boehringer Ingelheim Investigational Site, Kaunas
  - 1276.10.37004 Boehringer Ingelheim Investigational Site, Kaunas
  - 1276.10.37002 Boehringer Ingelheim Investigational Site, Klaipėda
  - 1276.10.37001 Boehringer Ingelheim Investigational Site, Vilnius
- Mexico (5):
  - 1276.10.52003 Boehringer Ingelheim Investigational Site, Durango
  - 1276.10.52001 Boehringer Ingelheim Investigational Site, Mexico City
  - 1276.10.52002 Boehringer Ingelheim Investigational Site, Mexico City
  - 1276.10.52005 Boehringer Ingelheim Investigational Site, Pachuca
  - 1276.10.52004 Boehringer Ingelheim Investigational Site, Tijuana
- New Zealand (2):
  - 1276.10.64001 Boehringer Ingelheim Investigational Site, Christchurch
  - 1276.10.64002 Boehringer Ingelheim Investigational Site, Greenlane East Auckland NZ
- Poland (7):
  - 1276.10.48001 Boehringer Ingelheim Investigational Site, Bialystok
  - 1276.10.48002 Boehringer Ingelheim Investigational Site, Bialystok
  - 1276.10.48008 Boehringer Ingelheim Investigational Site, Giżycko
  - 1276.10.48005 Boehringer Ingelheim Investigational Site, Katowice
  - 1276.10.48006 Boehringer Ingelheim Investigational Site, Katowice
  - 1276.10.48004 Boehringer Ingelheim Investigational Site, Krakow
  - 1276.10.48003 Boehringer Ingelheim Investigational Site, Warsaw
- Russia (8):
  - 1276.10.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1276.10.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 1276.10.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1276.10.70004 Boehringer Ingelheim Investigational Site, Moscow
  - 1276.10.70005 Boehringer Ingelheim Investigational Site, Moscow
  - 1276.10.70007 Boehringer Ingelheim Investigational Site, Moscow
  - 1276.10.70008 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1276.10.70009 Boehringer Ingelheim Investigational Site, Saint Petersburg
- South Africa (6):
  - 1276.10.27004 Boehringer Ingelheim Investigational Site, Paarl
  - 1276.10.27003 Boehringer Ingelheim Investigational Site, Parow
  - 1276.10.27006 Boehringer Ingelheim Investigational Site, Plumstead, Cape Town
  - 1276.10.27001 Boehringer Ingelheim Investigational Site, Pretoria
  - 1276.10.27005 Boehringer Ingelheim Investigational Site, Pretoria
  - 1276.10.27002 Boehringer Ingelheim Investigational Site, Somerset West
- Spain (6):
  - 1276.10.34005 Boehringer Ingelheim Investigational Site, Barcelona
  - 1276.10.34001 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1276.10.34003 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1276.10.34002 Boehringer Ingelheim Investigational Site, les Borges del Camp
  - 1276.10.34004 Boehringer Ingelheim Investigational Site, Sant Adria Del Besos
  - 1276.10.34006 Boehringer Ingelheim Investigational Site, Vic
- Ukraine (5):
  - 1276.10.38002 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1276.10.38007 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1276.10.38001 Boehringer Ingelheim Investigational Site, Kiev
  - 1276.10.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 1276.10.38005 Boehringer Ingelheim Investigational Site, Kyiv

REFERENCES:
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672

RESULTS

PARTICIPANT FLOW:
Groups:
- Empa 12.5mg BID: Oral administration of Empagliflozin (Empa) 12.5 mg twice daily (BID)
- Empa 25mg QD: Oral administration of Empagliflozin (Empa) 25 mg once daily (QD)
- Empa 5mg BID: Oral administration of Empagliflozin (Empa) 5 mg twice daily (BID)
- Empa 10mg QD: Oral administration of Empagliflozin (Empa) 10 mg once daily (QD)
- Placebo: Oral administration of Placebo tablets matching empagliflozin 25 mg, 10 mg, 5 mg, and 2.5 mg
Period: Overall Study
Arm/Group | Empa 12.5mg BID | Empa 25mg QD | Empa 5mg BID | Empa 10mg QD | Placebo
Started | 219 (randomised) | 218 (randomised) | 219 (randomised) | 220 (randomised) | 107 (randomised)
Completed | 205 | 205 | 202 | 201 | 103
Not Completed | 14 | 13 | 17 | 19 | 4
Not completed — Adverse Event | 5 | 5 | 4 | 13 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Non compliant with Protocol | 1 | 0 | 3 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 4 | 3 | 0
Not completed — Patient withdrawal (not due to AE) | 3 | 6 | 4 | 1 | 1
Not completed — For other reason | 4 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: FAS being defined as all patients randomised, treated with at least one dose of study drug, had a baseline Glycosylated Haemoglobin (HbA1c) and at least one on-treatment HbA1c assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empa 12.5mg BID | Empa 25mg QD | Empa 5mg BID | Empa 10mg QD | Placebo | Total
Number analyzed (Participants) | 215 | 214 | 215 | 214 | 107 | 965
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (9.9) | 58.2 (10.2) | 58.8 (9.8) | 58.5 (10.8) | 57.9 (11.2) | 58.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 100 | 95 | 106 | 52 | 445
  Male | 123 | 114 | 120 | 108 | 55 | 520

OUTCOME MEASURES:

1. Primary Outcome: HbA1c (Glycosylated Haemoglobin) Change From Baseline at Week 16
Description: Change from baseline in HbA1c (%) after 16 weeks of treatment. The term 'baseline' refers to the last observation prior to the first intake of any randomised study medication.
  Means provided are the adjusted means.
Time Frame: Baseline and 16 weeks
Population: Full Analysis Set (FAS) is the basis for the intention-to-treat analysis. FAS with last observation carried forward (LOCF) imputation is used as the primary method of accounting for missing data.
  Values after the patient started rescue medication were excluded from analysis (and imputed with an LOCF procedure).
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Empa 12.5mg BID | Empa 25mg QD | Empa 5mg BID | Empa 10mg QD | Placebo
Number analyzed (Participants) | 215 | 214 | 215 | 213 | 107
percentage of HbA1c | -0.83 (0.05) | -0.72 (0.05) | -0.66 (0.05) | -0.64 (0.05) | -0.22 (0.07)
Statistical Analysis 1: Comparison: Empa 5mg BID vs Empa 10mg QD; The primary objective was to test the non-inferiority of empagliflozin 5 mg BID versus empagliflozin 10 mg QD, and non-inferiority of empagliflozin 12.5 mg BID versus empagliflozin 25 mg QD, assuming a non-inferiority margin of 0.35%; Test type: Non-Inferiority or Equivalence — Null hypotheses for non-inferiority: H10: Mean change from baseline in HbA1c (%) after 16 weeks of treatment with empagliflozin 5 mg twice daily ≥ mean change from baseline in HbA1c (%) after 16 weeks of treatment with empagliflozin 10 mg once daily + 0.35% H20: Mean change from baseline in HbA1c (%) after 16 weeks of treatment with empagliflozin 12.5 mg twice daily ≥ mean change from baseline in HbA1c (%) after 16 weeks of treatment with empagliflozin 25 mg once daily + 0. 35%; p < 0.0001, ANCOVA — The two non-inferiority hypotheses H10 and H20 were tested using the Hochberg procedure in order to control the family-wise type I error at 0.025 (one-sided); ANCOVA: Treatment, geographical region, renal function (screening eGFR [MDRD] value)- fixed effects and baseline HbA1c- linear covariate; Adjusted mean difference = -0.02, 95% CI [-0.16 to 0.13], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Empa 12.5mg BID vs Empa 25mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.11, 95% CI [-0.26 to 0.03], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Empa 12.5mg BID vs Placebo; Superiority of once daily dose of empagliflozin (10 mg and 25 mg) versus placebo and superiority of twice daily dose of empagliflozin (5 mg and 12.5 mg) versus placebo in reducing HbA1c after 16 weeks of treatment was tested in an exploratory manner, to demonstrate assay sensitivity against placebo at 0.05 level (two-sided); Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.61, 95% CI [-0.79 to -0.44], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Empa 25mg QD vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.50, 95% CI [-0.68 to -0.32], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: Empa 5mg BID vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.44, 95% CI [-0.62 to -0.27], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Empa 10mg QD vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.42, 95% CI [-0.60 to -0.25], Standard Error of Mean 0.09

2. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline at Week 16
Description: Change from baseline in FPG (mg/dL) after 16 weeks of treatment. The term 'baseline' refers to the last observation prior to the first intake of any randomised study medication.
  Means provided are the adjusted means.
Time Frame: Baseline and 16 weeks
Population: FAS with LOCF has been used for FPG analyses
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Empa 12.5mg BID | Empa 25mg QD | Empa 5mg BID | Empa 10mg QD | Placebo
Number analyzed (Participants) | 213 | 214 | 213 | 213 | 107
mg/dL | -27.7 (2.0) | -22.7 (2.0) | -21.2 (2.0) | -17.6 (2.0) | -0.2 (2.8)
Statistical Analysis 1: Comparison: Empa 5mg BID vs Empa 10mg QD; Test type: Superiority or Other; ANCOVA; ANCOVA: Treatment, geographical region, renal function (screening (eGFR)[MDRD]value)-fixed effects and baseline HbA1c,baseline FPG-linear covariates; Adjusted mean difference = -3.6, 95% CI [-9.0 to 1.8], Standard Error of Mean 2.8
Statistical Analysis 2: Comparison: Empa 12.5mg BID vs Empa 25mg QD; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; Adjusted mean difference = -5.0, 95% CI [-10.4 to 0.5], Standard Error of Mean 2.8
Statistical Analysis 3: Comparison: Empa 12.5mg BID vs Placebo; Superiority of once daily dose of empagliflozin (10 mg and 25 mg) versus placebo and superiority of twice daily dose of empagliflozin (5 mg and 12.5 mg) versus placebo in reducing FPG after 16 weeks of treatment was tested in an exploratory manner, to demonstrate assay sensitivity against placebo at 0.05 level (two-sided); Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA:'Treatment','geographical region','renal function'(screening(eGFR)[MDRD]value)-fixed effects and 'baseline HbA1c',baseline FPG-linear covariate; Adjusted mean difference = -27.5, 95% CI [-34.2 to -20.9], Standard Error of Mean 3.4
Statistical Analysis 4: Comparison: Empa 25mg QD vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 3]; Adjusted mean difference = -22.5, 95% CI [-29.2 to -15.9], Standard Error of Mean 3.4
Statistical Analysis 5: Comparison: Empa 5mg BID vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 3]; Adjusted mean difference = -21.1, 95% CI [-27.7 to -14.4], Standard Error of Mean 3.4
Statistical Analysis 6: Comparison: Empa 10mg QD vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 3]; Adjusted mean difference = -17.5, 95% CI [-24.1 to -10.8], Standard Error of Mean 3.4

ADVERSE EVENTS:
Time Frame: 16 weeks + 1 week follow-up
Arm/Group | Empa 12.5mg BID | Empa 25mg QD | Empa 5mg BID | Empa 10mg QD | Placebo
Serious Adverse Events (participants affected / at risk) | 5/219 | 2/218 | 7/219 | 5/220 | 1/107
Other Adverse Events (participants affected / at risk) | 10/219 | 10/218 | 8/219 | 15/220 | 4/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empa 12.5mg BID (N=219) | Empa 25mg QD (N=218) | Empa 5mg BID (N=219) | Empa 10mg QD (N=220) | Placebo (N=107)
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Biliary adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Salivary gland pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa 12.5mg BID (N=219) | Empa 25mg QD (N=218) | Empa 5mg BID (N=219) | Empa 10mg QD (N=220) | Placebo (N=107)
Urinary tract infection (Infections and infestations) | 10 | 10 | 8 | 15 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.